CLINICAL TRIAL: NCT02976766
Title: Gypenosides Treatment for Optic Neuritis: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Gypenosides Treatment for Optic Neuritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrolment
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yi Du, Dr., First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GXON-001
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Optic Neuritis
Keywords: Neuroprotection; Clinical trial; Traditional Chinese medicine; Axonal loss; Jiaogulan; Gynostemma pentaphyllum; Optical coherence tomography
MeSH Terms: conditions — Optic Neuritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gypenosides (Experimental)
  Interventions: Drug: Gypenosides
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gypenosides — Participants will receive gypenosides 180 mg/day (60 mg three times a day) for 10 days.
  Other Names: Jiaogulan Zongdai
  Arms: Gypenosides
Drug: Placebo — Participants will receive placebo three times a day for 10 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether gypenosides are neuroprotective in patients with acute optic neuritis.

ELIGIBILITY:
Inclusion criteria

1. Male and female Chinese patients aged ≥18 to ≤60 years
2. Patients with a first episode of optic neuritis in the eye of interest
3. First symptoms of optic neuritis ≤28 days prior to the first administration of investigational product
4. Best corrected visual acuity in the eye of interest ≤0.8

Exclusion criteria

1. Pre-existing multiple sclerosis MS or NMO
2. Refractive media opacity
3. Hyperopia >5 diopters, myopia <-5 diopters, or astigmatism >3 diopters
4. Active tuberculosis, hepatitis, renal insufficiency, uncontrolled hypertension, diabetes mellitus, infection with HIV or syphilis, or any other conditions potentially interfering treatment trial
5. Other autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, etc)
6. Existing other retina or optic nerve diseases
7. Pregnant or females who plan to be pregnant during study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mean retinal nerve fibre layer thickness | 6 months

SECONDARY OUTCOMES:
Total macular volume | 6 months
Best corrected visual acuity | 6 months
Latency and amplitude of visual evoked potentials | 6 months
Mean visual field defect | 6 months
Number of participants with Adverse events | Screening until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Yi Du, MD, Principal Investigator — The First Affiliated Hospital of Guangxi Medical University, China
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China